CLINICAL TRIAL: NCT00259584
Title: A Prospective Longitudinal Study of the Management and Outcome of Superior Vena Caval Obstruction (SVCO)
Brief Title: Superior Vena Caval Obstruction (SVCO) - Management and Outcome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 01-0770-C
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2010-08

CONDITIONS: Superior Vena Cava Syndrome
MeSH Terms: conditions — Superior Vena Cava Syndrome | interventions — Therapeutics

INTERVENTIONS:
Behavioral: Management and Outcome of SVCO

SUMMARY:
All patients with symptomatic malignant SVCO deemed suitable for treatment either with radiation therapy or by stenting will be eligible. They will receive whichever treatment is deemed most clinically appropriate. Symptomatic response, time to onset of palliation, duration of symptom control and survival will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic clinical and radiological diagnosis of superior vena caval obstruction.
* Underlying histological diagnosis deemed appropriate for palliative radiotherapy as treatment by investigator. Patients with chemosensitive tumours such as small cell lung cancer (both untreated and recurrent), lymphoma and testicular tumours, will be eligible if radiation is deemed to be appropriate treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2001-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Improvement in an index symptom at 4 weeks as recorded by a daily symptom diary

SECONDARY OUTCOMES:
Time to onset of palliation
Duration of symptom control
Survival
Number of days spent in hospital
Requirement for further treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bezjak, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- University Health Network, Toronto, Ontario, Canada